CLINICAL TRIAL: NCT07205224
Title: Effects of Spinal Versus General Anesthesia on Perioperative Inflammatory Response in Percutaneous Nephrolithotomy (PCNL): The Role of Neutrophil-to-Lymphocyte Ratio (NLR), Red Cell Distribution Width (RDW), and Lactate-to-Albumin Ratio (LAR)
Brief Title: Inflammatory Response Under Spinal vs General Anesthesia in PCNL: NLR, RDW, LAR.
Acronym: SAGEPCNL
Status: Completed | Type: Observational
Sponsor: Sevim Şenol Karataş (Other)
Responsible Party: Sponsor-Investigator, Sevim Şenol Karataş, Principal Investigator,, Elazıg Fethi Sekin Sehir Hastanesi
Organization: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Other Study IDs: EFSH-ANES-2025-09-PERCUTANE
Record Dates: First submitted 2025-09-22; First posted 2025-10-03 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Nephrolithiasis; Postoperative Inflammation
Keywords: Percutaneous Nephrolithotomy; PCNL; Spinal Anesthesia; General Anesthesia; Inflammatory Response; Neutrophil-to-Lymphocyte Ratio (NLR); Red Cell Distribution Width (RDW); Lactate-to-Albumin Ratio (LAR)
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal Anesthesia Cohort: Adult patients (≥18 years, ASA I-III) undergoing percutaneous nephrolithotomy (PCNL) under spinal anesthesia. Routine perioperative laboratory values (NLR, RDW, LAR) will be recorded preoperatively and postoperatively.
  Interventions: Other: Anesthesia Type
- General Anesthesia Cohort: Adult patients (≥18 years, ASA I-III) undergoing percutaneous nephrolithotomy (PCNL) under general anesthesia. Routine perioperative laboratory values (NLR, RDW, LAR) will be recorded preoperatively and postoperatively.
  Interventions: Other: Anesthesia Type

INTERVENTIONS:
Other: Anesthesia Type — Patients receive either spinal or general anesthesia according to routine clinical decision-making. No investigational drug or device is administered.

SUMMARY:
This observational study compares the effects of spinal versus general anesthesia on the perioperative systemic inflammatory response in adults undergoing PCNL. Routine clinical laboratory values (NLR, RDW, LAR) obtained preoperatively and postoperatively will be recorded to evaluate between-group and within-group changes. No additional blood sampling will be performed beyond standard care.

DETAILED DESCRIPTION:
The study will be conducted at the Department of Anesthesiology and Reanimation, Elazığ Fethi Sekin City Hospital, among adult patients scheduled for PCNL (ASA I-III). The anesthesia type (spinal vs general) is determined by clinical requirements; investigators do not influence this choice.

Sampling windows:

Preoperative: within ≤6 hours before surgery

Postoperative: first sample obtained within 6-24 hours after surgery Parameters: NLR (neutrophil/lymphocyte), RDW, LAR; plus age, sex, ASA class, operative time, and in-hospital complications.

Statistics: Normality testing; between-group comparisons by independent t-test or Mann-Whitney U; within-group by paired t-test or Wilcoxon; categorical by chi-square; p<0.05 significant. Power considerations target ≥45 per group (total ≥90). No extra biospecimens will be collected beyond routine care.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years

ASA physical status I-III

Scheduled for percutaneous nephrolithotomy (PCNL)

Provided informed consent

Exclusion Criteria:

Active infection or sepsis

Known malignancy

Chronic inflammatory or autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus)

Current immunosuppressive therapy

Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years, ASA I-III) scheduled for percutaneous nephrolithotomy (PCNL) at a single tertiary care center. Eligible patients will be assigned to spinal or general anesthesia groups based on routine clinical decision-making. Routine perioperative laboratory values (NLR, RDW, LAR) will be collected preoperatively and postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Change in Neutrophil-to-Lymphocyte Ratio (ΔNLR) | Baseline (≤6 hours preoperative) and 24 hours postoperatively
  Difference in neutrophil-to-lymphocyte ratio (NLR) between preoperative (≤6 hours before surgery) and postoperative (6-24 hours after surgery) blood samples in spinal vs general anesthesia groups.

SECONDARY OUTCOMES:
Change in Red Cell Distribution Width (ΔRDW) | Baseline (≤6 hours preoperative) and 24 hours postoperatively
  Difference in RDW values between preoperative (≤6 hours before surgery) and postoperative (6-24 hours after surgery) blood samples in spinal vs general anesthesia groups.
Change in Lactate-to-Albumin Ratio (ΔLAR) | aseline (≤6 hours preoperative) and 24 hours postoperatively
  Difference in LAR values between preoperative (≤6 hours before surgery) and postoperative (6-24 hours after surgery) blood samples in spinal vs general anesthesia groups.
Postoperative Complications | From surgery until hospital discharge (up to 7 days)
  Occurrence of any PCNL-related complications (e.g., bleeding, infection) during index hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Şenol Karataş, Principal Investigator — Elazığ Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study uses routine clinical laboratory results and institutional restrictions do not allow sharing of raw patient-level data. Only de-identified aggregate results will be published in peer-reviewed journals upon request.

REFERENCES:
- [Background] Sankar K, Anand K, Ramani S, Gayathri B. A Randomized Control Trial to Compare Hemodynamic Parameters of Patients Undergoing Percutaneous Nephrolithotomy Under Combined Spinal-Epidural and General Anesthesia in a Tertiary Hospital. Local Reg Anesth. 2023 May 18;16:41-49. doi: 10.2147/LRA.S410510. eCollection 2023. PMID 37223489
- [Background] Wongyingsinn M, Kohmongkoludom P, Trakarnsanga A, Horthongkham N. Postoperative clinical outcomes and inflammatory markers after inguinal hernia repair using local, spinal, or general anesthesia: A randomized controlled trial. PLoS One. 2020 Nov 30;15(11):e0242925. doi: 10.1371/journal.pone.0242925. eCollection 2020. PMID 33253306
- [Background] Indra Rachman R, Birowo P, Nurullah G, Cho PSY, Atmoko W, Widyahening IS, Rasyid N. General versus spinal anesthesia in percutaneous nephrolithotomy: A systematic review and meta-analysis. F1000Res. 2023 Nov 1;12:281. doi: 10.12688/f1000research.124704.2. eCollection 2023. PMID 38618023
- See also: Elazığ Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation — https://elazigsehir.saglik.gov.tr/